CLINICAL TRIAL: NCT06516315
Title: Feasibility Study of an Angiographic Quantitative Flow Ratio-guided Endovascular Procedure in Patients With Lower Limbs Peripheral Arterial Disease.
Acronym: QFR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Medis Medical Imaging Systems B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 684_QFR; 2024-A00022-45 (Other: ANSM)
Record Dates: First submitted 2024-07-10; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Lower Limbs Peripheral Arterial Disease
Keywords: Lower Limbs Peripheral Arterial Disease; endovascular procedure; angiographic Quantitative Flow Ratio

STUDY DESIGN:
Intervention Model Description: Prospective feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- qfr (Experimental): Patients with indication for endovascular revascularization of a short stenosis of the superficial femoral artery (TASC A, Rutherford stage 2 to 6) :
  * Preoperative ultrasound, performed the day before or the day of surgery
  * Intraoperative angiography performed immediately prior to revascularization (routine care procedure whose duration is extended by research)
  * Quantitative analysis of angiography images will be performed post-procedure using Medis QFR®2.2 software.
  Interventions: Procedure: Preoperative ultrasound examination.; Procedure: Peroperatoire angiography procedure and QFR analysis

INTERVENTIONS:
Procedure: Preoperative ultrasound examination. — Preoperative ultrasound examination performed the day before or the day of surgery.
Procedure: Peroperatoire angiography procedure and QFR analysis — Intraoperative angiography will be performed immediately prior to revascularization. Quantitative analysis of angiography images will be performed post-procedure using Medis QFR®2.2 software.

SUMMARY:
The main objective of this study is to explore the feasibility of using the angiographic Quantitative Flow Ratio (QFR) as a tool to predict the success rate of endovascular revascularization in patients with superficial artery disease.

This is a prospective feasibility study. We aim to include 35 patients with indication for endovascular revascularization of a short stenosis of the superficial femoral artery. Intraoperative angiography will be performed immediately prior to revascularization. Quantitative analysis of angiography images will be performed post-procedure using Medis QFR®2.2 software.

DETAILED DESCRIPTION:
Approximately 202 million people are affected with lower extremity artery disease (LEAD) worldwide, of whom almost 40 million are living in Europe. LEAD usually appears after the age of 50 years, with an exponential increase after the age of 65. This rate reaches around 20% by the age of 80. In most studies, the proportion of symptomatic LEAD is 1:3 to 1:5 of all LEA.

The global burden of LEAD is considerable. In 2010, the years of life lost due to LEAD were estimated at 31.7, 15.1, and 3.7 years per 100,000 inhabitants in Western, Central, and Eastern Europe, respectively.

During the two last decade, indications of endovascular approach of femoropopliteal lesions have dramatically increased, to become the gold standard with a first endo strategy approach. In 2000, endovascular treatment was recommended for stenosis ≤ 5cm or occlusions ≤ 3cm. Today, the guidelines suggest endo approach for lesion until 25 cm In 2019, in France, 50 000 patients underwent an endovascular femoral popliteal revascularization, and drug eluting devices (Stents or Balloons). According to the Excellence in Peripheral Artery Disease Registry, early stent occlusion is about 5% during the 6 first months after procedure. Success rate of endovascular procedure is high, but many thrombosis are due to incomplete endovascular treatment, leading to early re-occlusion. Usually, quality and success assessment are made by the operator, based on images provided by a single plan angiography. Vascular surgeons face a lack of devices helping us to appreciate the quality of our revascularization per procedure. Endovascular ultrasounds (IVUS) or Optical Coherence Tomography(OCT) are not reimbursed in many countries. These devices are quite expensive and, like the FFR, require the introduction of dedicated devices into the arteries, thus increasing procedure's duration.

Similar situation can be seen in patients undergoing coronary percutaneous coronary intervention (PCI), current evidence indicates post-PCI suboptimal results. However, the combination of quantitative vessel analysis (QVA) with angiography-derived fractional flow reserve (FFR) assessment has shown promising improvements in PCI outcomes. A notable non-invasive solution for angiography derived FFR is Quantitative Flow Ratio (QFR), which includes quantitative vessel analysis (QVA) reporting significant enhancement in revascularization therapy.

Extending its potential benefits, QFR emerges as a non-invasive and cost-effective solution to improve revascularization outcomes for lower extremities.

MAIN OBJECTIVE The main objective of this study is to explore the feasibility of using QFR as a tool to predict the success rate of endovascular revascularization in patients with superficial artery disease.

METHODS:

1. Study design and Population This is a prospective feasibility study. We aim to include 35 patients with indication for endovascular revascularization of a short stenosis of the superficial femoral artery (TASC A, Rutherford stage 2 to 6). Intraoperative angiography will be performed immediately prior to revascularization. Quantitative analysis of angiography images will be performed post-procedure using Medis QFR®2.2 software.
2. Clinical variables:

   * Age
   * Sex
   * Height/Weight
   * Previous medical history
   * Rutherford classification
   * TASC lesion (only for sfa)
   * Procedure: - Type of treatment
   * Stents (type, length, diameter, number)
   * Amount of contrast
   * Xray duration
   * Xray Dose (Gy)
   * Technical success
   * Outcomes: 30 days patency
3. Angiography procedure and acquisition protocol Selective PCI will be performed using standard catheterization according to European society of Cardiology guidelines for lower extremity artery disease. At least two projections angles separated at least 25 degrees were acquired for the optimal view of the lesions. Details of the acquisition protocol are described in appendix B.
4. QCA and QFR analysis The 3D QCA and QFR analysis will be performed using a research version of software package QFR 2.2. QFR allows to match two diagnostic angiographic projections and create a 3D reconstruction of the interrogated vessel. From this reconstruction the following parameters will be derived: lesions length, QFR, delta(△) QFR, % diameter of stenosis, minimum lumen diameter, residual QFR, QFR pullback curve and derivative of QFR pullback curve (dQFR/ds).

ELIGIBILITY:
Inclusion Criteria:

* Patient with symptomatic Rutherford stage 2 to 6 AOMI with an indication for endovascular revascularization
* Patient with a simple lesion (TASC A) and short stenosis of the superficial femoral artery
* Patient affiliated to a health insurance system
* French-speaking patient
* Patient with free, informed and express oral consent

Exclusion Criteria:

* Renal failure patients with GFR < 30 ml/min
* Patient deprived of liberty
* Patients under court protection
* Pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-04-24 (Estimated); Study Completion 2025-05-24 (Estimated)

PRIMARY OUTCOMES:
Preoperative systolic velocity peak and intraoperative QFR | Day -1, Day 0
  Systolic velocity peak measured by preoperative ultrasound, performed the day before or the day of surgery, and QFR measured intraoperatively, immediately before the revascularization procedure.

SECONDARY OUTCOMES:
Percentage of stenosis | Day -1, Day 0
  Percentage of stenosis measured by preoperative ultrasound, performed the day before or the day of surgery.
Occurrence of a Major Adverse Limb Event (MALE) | Day 30
  Occurrence of a Major Adverse Limb Event (MALE) at 1 month post-op (D30): Acute ischemia OR Major amputation OR Re-intervention on revascularized limb (excluding minor amputation).
Re-hospitalization | Day 30
  Re-hospitalization for any reason at 1 month post-procedure (D30).
Revascularization | Day 30
  Revascularization (endovascular or surgical) of the treated area (Target Lesion Revascularization (TLR)) defined by re-intervention on the target lesion, including 1 cm above and below the target lesion.
Rutherford classification | Day 30
  Rutherford classification at 1 month post-op.
Dosimetry and dose of contrast medium | Day 0
  Dosimetry and dose of contrast medium injected during the procedure (D0).
Procedure envisaged by surgeon | Day 0
  Procedure envisaged by surgeon 1 and procedure envisaged by surgeon 2 after reading the QFR.
Creatinine levels and glomerular filtration rate | Day 5, Day 30
  Preoperative (D0) and postoperative (D5 and D30) creatinine levels and glomerular filtration rate.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime RAUX, Principal investigator, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Hôpital Paris Saint-Joseph - 185 Rue Raymond Losserand, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No